CLINICAL TRIAL: NCT01780467
Title: Role of Dopamine on Loss Aversion Behaviour: Study on Parkinsonian Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-0139; 2012-002768-28
Record Dates: First submitted 2013-01-21; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease
Keywords: Loss aversion; Dopamine; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

ARMS (2):
- patients with and without treatment by L dopa) (Experimental): to study the role of dopamine in the loss aversion phenomenon by comparing brain activity in parkinsonian patient with and without treatment with L Dopa, when they are exposed to mixed (gain/loss) gambles using money.
  Interventions: Behavioral: Role of dopamine
- healthy paired control (Other): to highlight the role of a dopamine depletion by comparing patient without treatment vs healthy paired control.
  Interventions: Behavioral: Role of dopamine

INTERVENTIONS:
Behavioral: Role of dopamine

SUMMARY:
Use lay language.

Many decisions involve the possibility of gaining or losing relative to the status quo. The loss aversion behaviour is a cognitive concept explaining that people are more sensitive to the possibility of losing objects or money than they are to the possibility of gaining the same objects or amounts of money.

We hypothesised that dopamine could be involved in the loss aversion behaviour. To highlight this, we have chosen a model of dopaminergic depletion : the Parkinson's disease The primary purpose of this protocol is to study the role of dopamine in the loss aversion phenomenon by comparing brain activity in parkinsonian patient with and without treatment with L Dopa, when they are exposed to mixed (gain/loss) gambles using money.

The second purpose is to highlight the role of a dopamine depletion by comparing patient without treatment vs healthy paired control.

2 groups :

* 20 parkinsonian patients (tested two times : with and without treatment by L dopa)
* 20 healthy paired control

Description of the protocol for patients :

J0 : Inclusion visit (duration : 4h):

* motor assessment (UPDRS)
* neuropsychological and psychiatric assessment (MMS, MATTIS, BREF, Stroop, Ardouin scale, UPPS, MADRS, Hamilton, LARS).

J0+1 day and J0 +2 days : 2 visits of MRI (magnetic resonance imaging) acquisition (with or without treatment) :

Each acquisition was composed by an orientation sequence+ an anatomic sequence + a functional sequence.

For healthy subjects, they have only one visit of 2 hours including a MMS, a MADRS and the MRI acquisitions.

DETAILED DESCRIPTION:
Use lay language.

Many decisions involve the possibility of gaining or losing relative to the status quo. The loss aversion behaviour is a cognitive concept explaining that people are more sensitive to the possibility of losing objects or money than they are to the possibility of gaining the same objects or amounts of money.

We hypothesised that dopamine could be involved in the loss aversion behaviour. To highlight this, we have chosen a model of dopaminergic depletion : the Parkinson's disease The primary purpose of this protocol is to study the role of dopamine in the loss aversion phenomenon by comparing brain activity in parkinsonian patient with and without treatment with L Dopa, when they are exposed to mixed (gain/loss) gambles using money.

The second purpose is to highlight the role of a dopamine depletion by comparing patient without treatment vs healthy paired control.

2 groups :

* 20 parkinsonian patients (tested two times : with and without treatment by L dopa)
* 20 healthy paired control

Description of the protocol for patients :

J0 : Inclusion visit (duration : 4h):

* motor assessment (UPDRS)
* neuropsychological and psychiatric assessment (MMS, MATTIS, BREF, Stroop, Ardouin scale, UPPS, MADRS, Hamilton, LARS).

J0+1 day and J0 +2 days : 2 visits of MRI (magnetic resonance imaging) acquisition (with or without treatment) :

Each acquisition was composed by an orientation sequence+ an anatomic sequence + a functional sequence.

For healthy subjects, they have only one visit of 2 hours including a MMS, a MADRS and the MRI acquisitions.

ELIGIBILITY:
Inclusion Criteria:

* Patients :
* Men or women aged between 35 -75 years
* Patients with an idiopathic Parkinson's disease according to UKPDSBB criterias with a disease evolution duration : 5-10 years)
* With fluctuations in end of doses + morning akinesia.
* Non dement (MMS>24 ; Mattis > 130)
* Affiliated to National Health system
* Having given their informed consent

Healthy controls

* Men or women aged between 35 to 75 years
* Non dement (MMS>24 )
* Affiliated to National Health system
* Having given their informed consent

Exclusion Criteria:

* Patients :
* Patients suffering of an atypical Parkinson syndrome
* Psychiatric pathology
* Tremor form (≥ 3 (item tremor of UPDRS))
* Patients with Impulsive control disorders
* Depression, dementia
* Pregnant
* Under guardianship
* In excluding period for another study
* Any contra-indication to MRI

Healthy subject

* Subject with neurological, psychiatric diseases
* Depression, dementia
* Pregnant
* Under guardianship
* In excluding period for another study
* Any contra-indication to MRI

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
percentage of signal modification | From day 1 (without L Dopa) to day 2 (with L Dopa)

SECONDARY OUTCOMES:
Cluster activation size | from day 1 (without L Dopa) to day 2 (with LDopa)
Brain activity indicators | from day 1 (without L Dopa) to day 2 (with L Dopa)

CONTACTS AND LOCATIONS:
Overall Officials: Ulla MIGUEL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France